CLINICAL TRIAL: NCT04906733
Title: Patient-derived Organoids of RAS/RAF Wild-type Metastatic Right Colon Cancer to Test the Sensitivity and Clinical Consistency of Combined Treatment of Cetuximab.
Brief Title: Cetuximab Sensitivity Correlation Between Patient-Derived Organoids and Clinical Response in Colon Cancer Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D1 Medical Technology (Shanghai) Co., Ltd, China (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: D1med-ZL01
Record Dates: First submitted 2021-05-27; First posted 2021-05-28 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Colon Cancer; Organoids; Metastatic Cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples of biopsy tissue from enrolled RAS/RAF wild-type metastatic right colon cancer patients are to be collected and subject to organoid isolation followed by the ex vivo drug sensitivity test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cancer patient: RAS/RAF wild-type metastatic right colon cancer patients receiving chemotherapy or chemotherapy combined target therapy treatment.
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor biopsy — Patients with RAS/RAF wild-type metastatic right colon cancer will receive biopsy before the standard treatment of chemotherapy or target therapy.

SUMMARY:
Eighty patients with RAS/RAF wild-type metastatic right colon cancer will be enrolled and undergo a fresh biopsy of tumor lesion before the standard treatment of chemotherapy. The investigators will establish organoids from the pre-treatment biopsies. Organoids will be exposed to the chemotherapy drugs or chemotherapy drugs combined with cetuximab used for each patient. The sensitivity of chemotherapy drugs or combined cetuximab will be tested in the organoids model. Chemotherapy strategies including 5-fluorouracil only, irinotecan only, oxaliplatin only, FOLFOX, and FOLFIRI. The purpose of this study is to evaluate the consistency and accuracy of a Patient-Derived Organoid (PDO) model of colon cancer to predict the clinical efficacy of combined treatment of cetuximab, which to formulate the best therapy regimen for each given patient.

DETAILED DESCRIPTION:
Investigators hypothesize that the cetuximab sensitivity test results on patient-derived organoids can be used to predict the treatment selection of patients with RAS/RAF wild-type metastatic right colon cancer.

Objectives

1. To assess the effective rate of cetuximab target therapy on RAS/RAF wild-type right colon cancer
2. To assess the consistency of organoid chemotherapy sensitivity and clinical chemotherapy efficacy
3. To assess the consistency of organoid cetuximab sensitivity and clinical cetuximab efficacy

The following points will be addressed:

1. The biopsy tissue of RAS/RAF wild-type metastatic right colon cancer will be collected and subject to ex vivo 3-D culture to establish patient-derived tumor organoids, which will be used for the drug sensitivity test.
2. Enrolled patients will treat with chemotherapy or chemotherapy combined target therapy. The medication regime and treatment cycle will be decided based on the clinical guideline and evidence-based medicine.
3. The patient-derived organoid-based drug sensitivity test will compare with clinical treatment data of chemotherapy or chemotherapy combined target therapy, followed by correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70 years old, no gender limit
2. The primary tumor is located in the right colon, including the ileocecal area, ascending colon, liver flexure, and the right part of the transverse colon.
3. Pathologically proved primary intestinal tumor with simultaneous / metachronous metastasis
4. Molecular pathology confirmed as RAS/RAF wild type
5. Can tolerate and cooperate with the completion of chemotherapy and targeted therapy
6. Tissues can be obtained through puncture or colonoscopy for organoid culture
7. Complete clinical data, as well as efficacy evaluation data, can be obtained

Exclusion Criteria:

1. Less than 18 years of age or more than 70 years of age
2. The primary tumor is located in the left colon or rectum
3. Pathology results can't confirm as colon cancer
4. RAS and RAF are mutant confirmed by molecular pathology
5. Refuse to cooperate and complete the treatment, or there is a contraindication for chemotherapy or targeted therapy
6. No available metastatic lesions tissue
7. Unable to obtain complete clinical data or efficacy evaluation data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Department of Colorectal Surgery in Fudan University Cancer Hospital is one of the largest colorectal cancer diagnosis and treatment centers in China. In 2019, more than 1,000 cases of recurrent and metastatic colorectal cancer were diagnosed and treated. It is sufficient to obtain samples for this study from patients diagnosed and treated in this department.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of ex vivo sensitivity test on patient-derived organoid models with clinical outcomes | 2021.05-2023.05
  The drug sensitivity tests on patient-derived tumor organoids will compare with the clinical response of the chemo- or targeted therapy treatment. The correlation of organoids sensitivity and patient response will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Peng, Dr., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04906733/ICF_000.pdf